CLINICAL TRIAL: NCT01754467
Title: NEAT! Technology to Increase Breaks in Sedentary Behavior in Adults With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Christine Pellegrini, Research Assistant Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CCDTR01
Record Dates: First submitted 2012-12-13; First posted 2012-12-21 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NEAT! (Experimental): Participants will use the NEAT! smartphone application and accelerometer over a 1 month period.
  Interventions: Behavioral: NEAT!

INTERVENTIONS:
Behavioral: NEAT! — Participants will wear the accelerometer and use the NEAT! application during waking hours for 1 month. The NEAT! app will prompt participants to stand up when they have been sitting for a prolonged period.

SUMMARY:
Sedentary behavior is associated with an increased risk of mortality and many health conditions including type 2 diabetes, obesity, cardiovascular disease, and metabolic syndrome, independent of the time spent in moderate-to-vigorous intensity physical activity (MVPA). Furthermore, independent of total sedentary time and MVPA, Healy et al. observed that individuals who had more breaks in sedentary time had lower 2-h plasma glucose. Recent experimental findings also suggests that breaking up prolonged bouts of sedentary behavior (≥ 20 minutes) with either light or moderate intensity activity for 2 minutes reduces postprandial glucose and insulin responses.10 Replacing sedentary time with light-intensity activity or nonexercise activity thermogenesis (NEAT) may help to reduce the health consequences of sedentary behavior. The purpose of this study is to develop a smartphone application (NEAT!) to encourage sedentary adults with diabetes to increase breaks in prolonged bouts of sedentary behavior objectively measured by an accelerometer. NEAT! will be refined by modifying technology created for the ENGAGED trial (RC1DK087126) and will work in conjunction with a Bluetooth enabled accelerometer that can detect bouts of sedentary behavior. When a sedentary bout (≥ 20 minutes) is detected, the smartphone application will trigger a reminder prompt to the user encouraging him/her to participate in NEAT for at least 2 minutes. Following the development, testing, and refining of the application, a sample of 10 sedentary adults with type 2 diabetes will be recruited to participate in a one month trial to examine the feasibility and acceptability of NEAT!. To our knowledge, this is the first study to design and examine the acceptability of a smartphone application that will target interrupting sedentary behavior with NEAT using objectively measured sedentary time in a diabetic population.

ELIGIBILITY:
Inclusion Criteria:

* 21-70 years of age
* have physician diagnosed type 2 diabetes that is currently being treated by dietary modification, oral agents, or insulin
* currently and plan on having an Android smartphone for the next 2 months
* be willing to wear an accelerometer and use the NEAT! application
* spend the majority of the day sitting.

Exclusion Criteria:

* unable to ambulate without assistance

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Pellegrini, Ph.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were only excluded if they did not meet the eligibility criteria or were no longer interested in participating.
Period: Overall Study
Arm/Group | NEAT!
Started | 9
Completed | 8
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | NEAT!
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 37.4 (9.9)

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of NEAT!
Description: How many participants would continue to use or use NEAT! in the future
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | NEAT!
Number analyzed (Participants) | 8
Participants | 7

2. Secondary Outcome: Adherence to NEAT!
Description: NEAT usage (days/month)
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: days
Arm/Group | NEAT!
Number analyzed (Participants) | 8
days | 21.9 (8.0)

3. Secondary Outcome: Breaks in Sedentary Behavior
Description: Changes in the number of breaks in sedentary behavior will be assessed via accelerometry between baseline and 1 month
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: breaks/day
Arm/Group | NEAT!
Number analyzed (Participants) | 8
breaks/day | 67.6 (15.1)

4. Secondary Outcome: Changes in Total Sedentary Time
Description: Changes in total sedentary behavior will be assessed via accelerometry between baseline and 1 month
Time Frame: Baseline and 1 month
Population: One individual outlier showed opposite changes as compared with the other participants and was 2.1 standard deviations above the mean for change in percent of day spent in sedentary behavior; thus this individual was excluded from this analysis.
Measure: Mean (Standard Deviation); unit: percentage of day spent sedentary
Arm/Group | NEAT!
Number analyzed (Participants) | 7
percentage of day spent sedentary | -8.1 (4.5)

ADVERSE EVENTS:
Arm/Group | NEAT!
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes